CLINICAL TRIAL: NCT04369716
Title: A Randomized, Crossover Study to Assess the Impact of Fruit Juice, Fruit Juice With Pomace, or Whole Fruit on Glycemic Response
Brief Title: The Impact of Fruit Juice, Fruit Juice With Pomace, or Whole Fruit on Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1709
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Glycemic Response
Keywords: fiber; fruit; pomace; postprandial glycemia

STUDY DESIGN:
Intervention Model Description: Conducted in 2 separate phases (1 phase/fruit) with 3 visits/phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Whole fruit 1 (Active Comparator): Oranges
  Interventions: Other: Whole oranges
- Whole fruit 2 (Active Comparator): Apples
  Interventions: Other: Whole Apples
- Juice 1 + pomace (Experimental): Orange Juice + orange pomace
  Interventions: Other: Orange juice + orange pomace
- Juice 2 + pomace (Experimental): Apple Juice + apple pomace
  Interventions: Other: Apple juice + apple pomace
- Juice 1 alone (Active Comparator): Orange Juice
  Interventions: Other: Orange juice
- Juice 2 alone (Active Comparator): Apple Juice
  Interventions: Other: Apple juice

INTERVENTIONS:
Other: Whole oranges — Navel oranges (227 g total)
  Arms: Whole fruit 1
Other: Whole Apples — Red Delicious apple with skin (230 g)
  Arms: Whole fruit 2
Other: Orange juice + orange pomace — Orange Juice (149 g) + orange pomace (100g) [40% pomace by weight]
  Arms: Juice 1 + pomace
Other: Apple juice + apple pomace — Apple Juice (129 g) + apple pomace (106 g) [45% pomace by weight]
  Arms: Juice 2 + pomace
Other: Orange juice — Orange Juice (250 g)
  Arms: Juice 1 alone
Other: Apple juice — Apple Juice (235 g)
  Arms: Juice 2 alone

SUMMARY:
The primary aim of this clinical trial is to compare the effects of a whole orange, orange juice alone, and orange juice with pomace, and a whole apple, apple juice alone, apple juice with pomace on glycemic response. Fruit pomace is a fiber-rich byproduct that is isolated during normal juice production of fruits, such as orange and apple.

DETAILED DESCRIPTION:
Study products are matched on total sugar and fiber. Phase I consists of 3 orange study products and Phase II consists of 3 apple study products. Subjects consume one fruit test portion or beverage test portion per visit day with at least a 3 day washout in between.

24 hr diet records are reviewed each test day to verify food and drink consistency and a diet containing at least 150 g of carbohydrate. Subjects arrive fasted (10-14 h, water only), are asked to maintain adequate hydration; and refrain from vigorous physical activity (24 h), alcohol consumption (24 h), and tobacco products (for at least 1 h).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a generally healthy male or female, 18-65 years of age, inclusive.
2. Subject has a BMI of 18.5 to 29.9 kg/m2, inclusive, at Visit 1.
3. Subject has a rating of 7 to 10 on the Vein Access Scale at Visit 1.
4. If a smoker, subject has no plans to change smoking habits during the study period and is able to abstain from tobacco products at least 1 h prior to and during each test visit
5. Subject is on a stable dose of vitamins, minerals, and other supplements throughout the trial and is willing to maintain the current use throughout the trial. On test days, subject agrees not to take any vitamins, minerals, or other dietary supplements until dismissal from the clinic. Failure to comply will result in a rescheduled test visit.
6. If a female on oral contraceptives, the subject must be on a stable dose of oral contraceptives [defined as same dose for the past 90 d
7. If applicable, subject must be on a stable dose of.osteoporosis medication, anti-hypertensive medication, aspirin, and/or thyroid medication.
8. Subject is normally active and judged by the Investigator to be in general good health on the basis of medical history.
9. Subject is willing to maintain physical activity patterns, body weight, and habitual diet throughout the trial.
10. Subject is willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to and during test visits.
11. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the Investigators.
12. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.

Exclusion Criteria:

1. Subject has diagnosed diabetes mellitus (Type 1 or Type 2) or fasting glucose ≥110 mg/dL at Visit 1. No retest allowed.
2. Subject has the presence of a gastrointestinal disease or condition that could potentially interfere with absorption of the study product (including but not limited to inflammatory bowel diseases, ulcers), including history of gastrointestinal surgery (e.g., for weight reduction).
3. Subject has a history or presence of clinically important endocrine, cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary (including uncontrolled asthma), hepatic, renal, hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), or biliary disorders, in the opinion of the Clinical Investigator.
4. Subject has a history of bariatric surgery.
5. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian), in the opinion of the Clinical Investigator.
6. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at Visit 1. One retest will be allowed.
7. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
8. Subject has experienced any major trauma or any other surgical event within three months
9. Subject has a known allergy, intolerances, or sensitivity to any of the ingredients in the study products.
10. Subject has had a weight loss or gain >4.5 kg in the 3 months prior to Visit 1.
11. Subject has any signs or symptoms of an active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved (at the discretion of the Investigator) and any treatment (e.g., antibiotic therapy) has been completed at least 5 d prior to testing.
12. Subject has a recent history of (within 12 months of Visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse define as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
13. Subject has used medications known to influence carbohydrate metabolism, including, but not limited to, protease inhibitors, antipsychotics, adrenergic receptor blockers, diuretics, anti-diabetic agents, and systemic corticosteroids, within 30 d of Visit 1.
14. Subject has used weight-loss drugs (including over-the-counter medications and/or supplements) or programs within 30 d prior to Visit 1.
15. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
16. Subject has been exposed to any non-registered drug product within 30 days prior to Visit 1.
17. Subject has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Positive incremental area under the curve (iAUC) for blood glucose | t = -15, -5, 15, 30, 45, 60, 90, and 120 min where t = 0 min is the start of study product consumption
  Blood serum

SECONDARY OUTCOMES:
iAUC0-120 min for insulin | t = -15, -5, 15, 30, 45, 60, 90, and 120 min where t = 0 min is the start of study product consumption
  Blood serum
Maximum concentration (Cmax) for blood glucose | t = -15, -5, 15, 30, 45, 60, 90, and 120 min where t = 0 min is the start of study product consumption
  Blood serum
Time to maximum concentration (tmax) for blood glucose | t = -15, -5, 15, 30, 45, 60, 90, and 120 min where t = 0 min is the start of study product consumption
  Blood serum
Maximum concentration (Cmax) for insulin | t = -15, -5, 15, 30, 45, 60, 90, and 120 min where t = 0 min is the start of study product consumption
  Blood serum
Time to maximum concentration (tmax) for insulin | t = -15, -5, 15, 30, 45, 60, 90, and 120 min where t = 0 min is the start of study product consumption
  Blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lawless, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- BioFortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No